CLINICAL TRIAL: NCT01093339
Title: To Determine if Sleep Deprivation Results in Increased Esophageal Acid Exposure, and if This Effect is Mediated in Gastroesophageal Reflux Disease (GERD)Patients by Altering Appetite Regulation
Brief Title: To Determine if Sleep Deprivation Results in Increased Esophageal Acid Exposure
Acronym: IRUSESOM0428
Status: Completed | Type: Observational
Sponsor: Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Ronnie Fass MD, SArizona VAHCS
Other Study IDs: SLEEP DEPRIVATION
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Gastroesophageal Disease
Keywords: GERD; SLEEP DEPRIVATION; APPETITE REGULATION; GHRELIN; LEPTIN
MeSH Terms: conditions — Gastroesophageal Reflux; Sleep Deprivation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples collected and stored -80 freezer in GI lab.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Subjects w/ condition and subjects w/o condition of GERD (gastroesophageal reflux disease)

SUMMARY:
The purpose of this study is to determine if sleep deprivation results in increased esophageal acid exposure in healthy controls and gastroesophageal reflux disease (GERD) patients.

DETAILED DESCRIPTION:
To determine if increased esophageal acid exposure is mediated by altering appetite regulation. To assess if there is any relationship between sleep deprivation and the serum level of TNF-alfa (a protein that can be elevated in inflammation).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female - 18-80
* 2 or more episodes of heartburn a week for last 3 months

Exclusion Criteria:

* Previous upper GI surgery
* Underlying co-morbidity
* Narcotic medications
* Psychotropic's and Benzodiazapines medications
* Hx of psychological abnormalities
* Hx of ETOH in previous 6 mos.
* Diabetes Mellitus
* Neuropathy
* Seizures
* Sleep Apnea
* Co-morbidity that interfere w/sleep
* Women who are pregnant, or childbearing yrs, not on BC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 subjects w/ GERD 25 subjects w/o GERD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — SArizona VAHCS
Locations (1):
- SArizonaVAHCS, Tucson, Arizona, United States